CLINICAL TRIAL: NCT00392418
Title: The Effectiveness of Flexible Administration of Sprinkles® in a Mixed Population of Anemic and Non-anemic Infants and Young Children in Rural Bangladesh.
Brief Title: Flexible Administration of Sprinkles® in Infants and Young Children in Rural Bangladesh.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Collaborators: Heinz Endowments (Other)
Responsible Party: Principal Investigator, Stanley Zlotkin, Chief, Global Child Health, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1000005427
Record Dates: First submitted 2006-10-24; First posted 2006-10-26 (Estimated); Last update posted 2021-04-19 (Actual); Status verified 2021-04

CONDITIONS: Anemia
Keywords: iron deficiency anemia; hematologic disease; infancy; pediatrics; Sprinkles®; iron; micronutrient
MeSH Terms: conditions — Anemia; Anemia, Iron-Deficiency; Hematologic Diseases | interventions — Iron

INTERVENTIONS:
Drug: Multiple micronutrient supplement (iron)

SUMMARY:
Millions of people worldwide are affected by iron deficiency anemia (IDA). IDA is a widespread serious public health problem, especially for infants in developing countries mainly because of inadequate intake of iron due to the poor bioavailability of dietary iron in predominately cereal based diets. One of the ways to combat iron deficiency anemia is by supplementation to targeted populations. Although iron drops have been used, they have been largely unsuccessful in reducing the prevalence of anemia because of compliance, distribution and supply issues. Sprinkles® are a new approach to iron delivery that is as efficacious as iron drops and more acceptable. For Sprinkles® to be implemented into nation-wide programs as a sustainable alternative to current iron supplementation approaches, an optimal model of use and distribution for Sprinkles® needs to be established. By comparing daily versus flexible use of Sprinkles® (60 sachets over 60, 90 and 120 days) among infants and young children aged 6-24 months, the primary objectives are to study the effect of the three administration models of Sprinkles® on changes in:

1. hemoglobin concentration; and
2. compliance or adherence to the intervention.

ii. The secondary objective of this study is to determine the acceptability of each of the three intervention models.

We hypothesize that adherence will be greater and hemoglobin concentration response will be higher in those given 'flexible' instructions to use all of the Sprinkles® supplied over a specific period of time compared to those given strict instructions for daily use.

DETAILED DESCRIPTION:
Study Design

This study will follow a community-based cluster randomized clinical trial design involving three intervention groups. Total number of villages included in the study will be determined by the availability of the eligible children. In each village, all eligible children will be screened through house-to-house visits. After the screening, all the children will be randomized by village using a table with randomly assorted table into one of three groups:

* Daily use of 60 Sprinkles® sachets over 60 days.
* Flexible use of 60 Sprinkles® sachets over 90 days.
* Flexible use of 60 Sprinkles® sachets over 120 days.

In all groups, assessments will be done at baseline, at the end of a group's intervention and at 6 months after intervention in each group for follow-up.

The study will take place in Kaligong sub-district in Bangladesh. All villages in Kaligonj sub-district consist of plain agricultural land. Subsistence farming is the major source of livelihood. Rice is the commonly eaten staple mixed with lentil and vegetable curry and occasionally with pieces of fish and meat. Similar to the rest of the plain areas of the country, malnutrition among women and children is widespread, but malaria is extremely uncommon and the prevalence of hookworm is fairly low (less than 2%%).

ELIGIBILITY:
Inclusion Criteria:

* Age 6-24 months.
* Hemoglobin concentration > =70 g/L.
* Consuming at least one regular meal of complementary food per day.
* Reportedly free from any acute or chronic illness.
* Permanent resident of the village.
* Not receiving any other form of iron supplementation.
* Parental consent obtained.

Exclusion Criteria:

* Severe anemia (hemoglobin concentration <70 g/L).

Ages: 6 Months to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 360
Dates: Start 2004-05; Study Completion 2005-03

PRIMARY OUTCOMES:
hemoglobin concentration | at end of treatment and 6 months post-treatment
adherence measured by the number of sachets used | end of treatment

SECONDARY OUTCOMES:
Acceptability measured through interview with mothers
weaning food practice at treatment end and 6 months post-treatment
length and weight at treatment end and 6 months post-treatment
morbidity from diarrhea and acute respiratory infections at treatment end and 6 months post treatment

CONTACTS AND LOCATIONS:
Overall Officials: Stanley H Zlotkin, PhD, Principal Investigator — The Hospital for Sick Children, Toronto, Canada
Locations (1):
- Research and Evaluation Division, BRAC, Dhaka, Bangladesh